CLINICAL TRIAL: NCT05247879
Title: Clinical Effectiveness and Safety of a Novel Oral Rehydration Solution in Children Ages 1-5 Years Presenting to Hospital With Mild or Moderate Dehydration Gastroenteritis: Randomized, Open-label, Controlled Trial
Brief Title: Clinical Effectiveness and Safety of a Novel Oral Rehydration Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5003
Record Dates: First submitted 2022-01-07; First posted 2022-02-21 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Gastroenteritis Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Commercial reduced-osmolarity oral rehydration solution (ORS (Active Comparator)
  Interventions: Dietary Supplement: Glucose containing Oral Rehydration Solution (ORS)
- VS011, new children's ORS, a sugar-free blend of amino acids and electrolytes (Experimental)
  Interventions: Dietary Supplement: Sugar free - amino acid and electrolyte ORS

INTERVENTIONS:
Dietary Supplement: Glucose containing Oral Rehydration Solution (ORS) — Oral rehydration solution
  Arms: Commercial reduced-osmolarity oral rehydration solution (ORS
Dietary Supplement: Sugar free - amino acid and electrolyte ORS — Glucose free oral rehydration solution
  Arms: VS011, new children's ORS, a sugar-free blend of amino acids and electrolytes

SUMMARY:
This is a randomised, controlled, open-label study to determine the clinical effectiveness and safety of a novel ORS compared with a commercial ORS in children 1 to 5 years of age attending emergency departments with gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* 1 to 5 years of age, inclusive at randomization
* Hospitalized with mild to moderate dehydration due to ongoing diarrhea
* Signed informed consent obtained for child's participation in the study

Exclusion Criteria:

* Severe dehydration and/or use of IV fluids for current hospitalization
* Experiencing bloody diarrhea or diarrhea due to Cholera, Dysentery, persistent/chronic diarrhea, diarrhea with severe malnutrition, diarrhea associated with recent antibiotic use
* In the opinion of the Investigator, not suitable for treatment with ORS
* Have any underlying disease or disorder that may, in the opinion of the Investigator, affect the results of the study if they were enrolled (includes, but is not limited to, gastrointestinal disorders such as Crohn's disease or other inflammatory bowel disease or congenital malabsorption disorders)
* Cause of the dehydration is something other than diarrhea
* Known to be allergic to any of the components of the Investigational ORS

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Clinically assessed adequate rehydration based on clinical judgement of change in or absence of presenting symptoms from baseline (i.e. heart rate, urine output, etc.) | every 4 hours up to 24 hours or hospital discharge, whichever occurs first
  Assess change in clinical hydration status from presenting baseline status

SECONDARY OUTCOMES:
Clinical Assessment of patient's hydration status based on presenting symptoms (i.e. heart rate, urine output, etc.) | Baseline
  5 point scale, 1(no discomfort) minimum, 5 (severe discomfort) maximum
Study ORS intake (units) | Every 4 hours up to 24 hours or hospital discharge, whichever occurs first
Use of IV fluids | up to 24 hours or hospital discharge, whichever occurs first
Weight | Every 4 hours up to 24 h or at hospital discharge, whichever occurs first
  kg
Participant comfort questionaire | baseline and 24 hours or hospital discharge, whichever occurs first
Parent satisfaction questionnaire | baseline and 24 hours or hospital discharge, whichever occurs first
Frequency of vomiting | every 4 hours up to 24 hours or hospital discharge, whichever occurs first
Frequency episodes of urination | every 4 hours up to 24 hours or hospital discharge, whichever occurs first
Frequency of liquid/watery stool | every 4 hours up to 24 hours or hospital discharge, whichever occurs first
Time to resolution of liquid/water stool | up to 24 hours or hospital discharge, whichever comes first
Stool for bacterial pathogen culture and viral antigens | up to 24 hours or hospital discharge, whichever comes first
Time ready for discharge | At discharge or 48 hours whichever occurs first
Medically confirmed adverse events collected throughout the study period | 0 hours through 7 days post discharge
Record patient use of antibiotics during hospitalization | up to 24 hours or hospital discharge, whichever comes first

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Naresuan University Hospital, Phitsanulok

IPD SHARING:
Plan to Share IPD: No